CLINICAL TRIAL: NCT06804005
Title: Effects of Mandala Coloring and Music Activity on Future Anxiety and Subjective Well-Being in Nursing Students: A Randomized Controlled Trial
Brief Title: Mandala Coloring, Music, and Nursing Students' Anxiety and Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Abdurrahim UYANIK, Lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Gaziosmanpasa-CBAU
Record Dates: First submitted 2025-01-13; First posted 2025-01-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Nursing Students; Well-being; Anxiety
Keywords: nursing student; well being; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized-controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Music group (Experimental): The music activity will be performed with the research applicant's instrument (guitar) after the repertoire list is created with the songs the students want. The music will be sung continuously in an area equipped with a sound system so that the subjects can listen comfortably without headphones, and will be performed with the participation of the students along with peer support. Each intervention activity will last approximately 60 minutes.
  Interventions: Behavioral: Music group
- Mandala coloring (Experimental): In the mandala coloring activity, they will be asked to choose the picture they want from the mandala coloring booklets and color it however they want. This activity will take approximately 60 minutes.
  Interventions: Behavioral: mandala group
- Control Group (No Intervention): They will only fill out survey forms.

INTERVENTIONS:
Behavioral: Music group — Music will be sung continuously in an area equipped with a sound system so that subjects can listen comfortably without headphones, and will be performed with the participation of students and peer support. Each intervention activity will last approximately 60 minutes.
  Arms: Music group
Behavioral: mandala group — In the mandala coloring activity, they will be asked to choose the picture they want from the mandala coloring booklets and color it however they want. This activity will take approximately 60 minutes.
  Arms: Mandala coloring

SUMMARY:
This study aims to examine the effects of creative approaches aimed at reducing anxiety and increasing happiness by addressing the future concerns and subjective well-being levels of university students. Although the negative effects of anxiety on students' academic and personal lives have been widely examined in the literature, studies on the effectiveness of artistic interventions such as mandala painting and music therapy in reducing anxiety are limited. In this context, the study aims to fill an important gap in the field by evaluating the combined effects of these two methods. In particular, it aims to provide evidence-based methods that will improve the mental and emotional states of university students with practical results, thus making a positive contribution to both individual health and educational processes.

Main Hypotheses of the Study:

* H1: There is a difference between the levels of future anxiety and subjective well-being between nursing students who painted mandalas and those who did not.
* H1-0: There is no difference between the levels of future anxiety and subjective well-being between nursing students who painted mandalas and those who did not.
* H2: There is a difference between the levels of future anxiety and subjective well-being between nursing students who participated in the music activity and those who did not.
* H2-0: There is no difference between the levels of future anxiety and subjective well-being between nursing students who participated in the music activity and those who did not.

Research Questions:

* Is mandala painting and music activity effective in reducing nursing students' future anxiety levels?
* Is mandala painting and music activity effective in increasing nursing students' subjective well-being levels?
* Which of the mandala painting and music activity applications is more effective on nursing students' future anxiety and subjective well-being?

DETAILED DESCRIPTION:
While performing mandala painting activities, individuals focus on the present moment, especially when the individual's attention is focused on the activity at hand, and therefore it is accepted that such artistic practices are based on awareness (Chen et al., 2024). Studies in the literature report that mandala painting is an effective method in reducing negative mood and anxiety (Babouchkina and Robbins, 2015; Stinley et al., 2015; Sandmire et al., 2016). Another method used to reduce anxiety is music activities. Music therapy is a field in which music and music-related activities are used to meet the physical, mental, social and psychological needs of individuals. It can be said that music appeals to people's emotions and thoughts with its unique language and forms of expression. Music, which is considered one of the oldest treatment methods in history, is widely used in different cultures. In addition, music has positive effects on the treatment of mental illnesses and on some hormones that regulate mood. Music interventions that are clinically and evidence-based within a therapeutic relationship to achieve individual-specific goals have led to music therapy being accepted as a scientific treatment method. Music can affect people's emotional state, lead to changes in their behaviors, create psychological and physiological effects, and facilitate communication, which emphasizes the importance of music as a therapeutic element (Bulfone et al., 2019; Şen, 2022). This research aims to examine the effects of creative approaches to reduce anxiety and increase happiness by addressing university students' future concerns and subjective well-being levels. Although the negative effects of anxiety on students' academic and personal lives have been widely examined in the literature, studies on the effectiveness of artistic interventions such as mandala painting and music therapy in reducing anxiety are limited. In this context, the research aims to fill an important gap in the field by evaluating the combined effect of these two methods. In particular, it aims to provide evidence-based methods that will improve the mental and emotional states of university students with its practical results, and to make a positive contribution to both individual health and educational processes. As a result, university students' concerns about the future can have negative effects on both their mental and physical health. In this context, strategies to reduce anxiety about the future and approaches to increase happiness will play an important role in improving students' general well-being. Artistic and musical activities can reduce anxiety by strengthening individuals' emotional and mental states and help them live a healthy life. Such activities not only contribute to the personal development of university students, but also provide important opportunities for them to serve society as more creative, productive and healthy individuals. In addition, research in this area will make a valuable contribution to the literature and create a wider impact.

Data Collection Tools

* Sociodemographic Characteristics Form: consists of 4 questions in total, including age, gender, class, and region of birth.
* Subjective Well-Being Scale: The scale developed by Tuzgöl- Dost (2005) consists of 46 items. The aim of the scale is to determine the subjective well-being levels of individuals by determining the frequency and intensity of positive and negative emotions they experience with their cognitive evaluations about their lives. The subjective well-being scale consists of personal judgments about living spaces and positive and negative emotional expressions. The response system is in the form of a five-point Likert scale for each expression as "(5) Completely Appropriate", "(4) Mostly Appropriate", "(3) Partially Appropriate", "(2) Somewhat Appropriate", (1) "Not Appropriate at All". 26 of the scale items are positive and 20 are negative. Negative expressions; These are items 2, 4, 6, 10, 13, 15, 17, 19, 21, 24, 26, 28, 30, 32, 35, 37, 38, 40, 43, and 45. Negative statements are scored by reversing the scores. Positive statements are items 1, 3, 5, 7, 8, 9, 11,12, 14, 16, 18, 20, 22, 23, 25, 27, 26, 29,31, 33, 34, 36, 39, 41, 42, and 44. The lowest score that can be obtained from the scale is 46 and the highest score is 230. A high score indicates a high level of subjective well-being. Cronbach's alpha internal consistency coefficient is 93, and the test-retest reliability coefficient is 86. Subjective well-being reliability coefficients show that the scale is suitable for measuring the subjective well-being levels of university students.
* Future Anxiety Scale in University Students: The 5-point Likert-type Future Anxiety Scale, consisting of a total of 19 items, was developed by Geylani and Yıldız in 2022. The first factor of the scale was called "Future Fear" and the second factor was called "Hopelessness about the Future". The internal consistency of the scale was evaluated with the item-total score correlation and Cronbach's α method. Cronbach's α values were calculated as 0.91 for the entire scale, 0.95 for the first factor, and 0.88 for the second factor (Geylani & Yıldız, 2022).

ELIGIBILITY:
Inclusion Criteria:

* Studying in the Nursing Department of Erbaa Faculty of Health Sciences
* Volunteering to participate in the study

Exclusion Criteria:

* Filling out scales and forms incompletely
* Wanting to leave the research
* Not participating fully in activities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Well-being | 4 weeks
  The Subjective Well-being Scale assesses individuals' cognitive evaluations of their lives and the frequency and intensity of positive and negative emotions they experience.

SECONDARY OUTCOMES:
Future Anxiety | 4 weeks
  Evaluates nursing students' fear of the future and hopelessness levels about the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR